CLINICAL TRIAL: NCT04935177
Title: An Open-label, Controlled, Randomized Phase 3 Trial Evaluating 12-month Kidney Function in Highly Sensitized (cPRA ≥99.9%) Kidney Tx Patients With Positive XM Against a Deceased Donor, Comparing Desensitization Using Imlifidase With SoC
Brief Title: Renal Function in Highly Sensitized Patients 1 Year After Desensitization With Imlifidase Prior to DD Kidney Tx
Acronym: ConfIdeS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-HMedIdeS-17
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplantation in Highly Sensitized Patients
Keywords: Desensitization; Highly sensitized; Positive crossmatch; Unlikely to be transplanted; Renal transplantation; Deceased donor
MeSH Terms: interventions — Mac-1-like protein, Streptococcus; Plasma Exchange; Immunoglobulins, Intravenous; Rituximab; eculizumab

STUDY DESIGN:
Intervention Model Description: Open-label, controlled and randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Imlifidase (Experimental): Imlifidase, is provided as a freeze-dried powder for concentrate for solution for infusion, 11 mg per vial. After reconstitution with sterile water for injection, the concentrate contains 10 mg/mL imlifidase. Imlifidase is administered intravenously as one infusion of 0.25 mg/kg over 15 minutes generally 24 hours prior to transplantation. A second dose of 0.25 mg/kg may be given if the first imlifidase dose is considered not to have had sufficient effect.
  Interventions: Drug: Imlifidase
- Best available treatment (Other): Institution-specific desensitization protocol (i.e. any combination of plasma exchange (PLEX), intravenous IVIg, anti-CD20 antibody, and eculizumab) where appropriate OR remain on wait list for a more compatible organ offer
  Interventions: Procedure: PLEX; Drug: IVIg; Drug: Anti-CD20 antibodies; Drug: Eculizumab; Other: Remain on wait list

INTERVENTIONS:
Drug: Imlifidase — Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly selective towards IgG. The cleavage of IgG generates one F(ab')2- and one homodimeric Fc-fragment and efficiently neutralizes Fc-mediated activities of IgG.
  Other Names: IdeS, HMED-IdeS
  Arms: Imlifidase
Procedure: PLEX — PLEX is performed according to the respective site's standard procedure for desensitization.
  Other Names: Plasma exchange, PE
  Arms: Best available treatment
Drug: IVIg — IVIg prepared from a pool of immunoglobulins from the plasma of thousands of healthy donors is administered in accordance with respective site's standard procedure for desensitization.
  Other Names: Intravenous immunoglobulin
  Arms: Best available treatment
Drug: Anti-CD20 antibodies — Rituximab and other anti-CD20 according to the respective site's standard procedure for desensitization.
  Other Names: Rituximab
  Arms: Best available treatment
Drug: Eculizumab — Eculizumab according to the respective site's standard procedure for desensitization.
  Other Names: Soliris
  Arms: Best available treatment
Other: Remain on wait list — Remain on wait list for a more compatible organ offer if desentization with institutional protocol is not appropriate
  Arms: Best available treatment

SUMMARY:
An open-label, controlled, randomized Phase 3 trial evaluating 12-month kidney function in highly sensitized (cPRA ≥99.9%) kidney transplant patients with positive crossmatch against a deceased donor, comparing desensitization using imlifidase with standard of care

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo pre-screening to determine eligibility for study entry.

Once an organ offer is received, a virtual crossmatch (vXM) is performed. If the crossmatch is considered predictive of a positive flow cytometry crossmatch (FCXM), the patient will be evaluated if eligible to receive the desensitization currently in use at the study site. Subsequently the patient will be randomized in a 1:1 ratio to the imlifidase or the control arm.

If the patient is randomized to the imlifidase arm, the organ will be accepted and shipped, and the patient will proceed to imlifidase treatment (generally within 24 h prior to transplantation) followed by transplantation. If the patient is randomized to the control arm, transplantation made possible by the local desensitization regimen will occur. If the institution-specific desensitization protocol is deemed not to be successful, the organ offer will be turned down, and the patient will remain active on the waiting list and remain in the trial, while the kidney will be allocated to another recipient through the kidney allocation system (KAS).

All transplanted patients will receive induction therapy and maintenance immunosuppression. All patients will be followed for 12 months.

Estimated glomerular filtration rate (eGFR) will be assessed 12 months after randomization as the primary endpoint reasonably likely to predict a clinical benefit in patient survival.

All patients with donor specific antibodies (DSA) are at risk of developing antibody-mediated rejection (AMR). Imlifidase removes DSA quickly and efficiently at the time of transplantation but, as with other desensitization methods, the antibodies are expected to re-occur after transplantation. In the imlifidase treatment arm, and for desensitized control arm patients, protocol kidney biopsies will be performed at the time of transplantation and at 1 year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent obtained before any trial-related procedures
* Male or female age 18-70 years at the time of screening
* Chronic kidney disease (CKD) stage 5, highly sensitized as evaluated by standard selection criteria, and active on the OPTN waiting list for a DD kidney transplant
* Original calculated panel reactive antibody (cPRA) ≥99.9%
* Virtual crossmatch (vXM), predictive of a positive crossmatch to an available deceased donor (DD)
* Willingness and ability to comply with the protocol
* Willingness to participate in the planned 4-year extension trial

Exclusion Criteria:

* High dose IVIg (2 g/kg) treatment within 28 days prior to imlifidase treatment
* Previous treatment with imlifidase
* Breast feeding or pregnancy
* Women of child-bearing potential not willing or able to practice FDA-approved forms of contraception, or abstinence. Two medically acceptable methods of highly effective contraception must be used for the duration of the study (e.g. oral, transdermal, intravaginal, injectable or implantable contraceptive; intrauterine device; intrauterine hormone-releasing system; vasectomized partner; bilateral tubal occlusion; or double barrier method). For a woman to be considered postmenopausal this ascertainment must be made according to medical records and clinical history and may be aided by measurement of elevated postmenopausal serum gonadotropin levels (FSH).
* ABO blood group incompatible transplantations (A2 or A2B kidneys will not be accepted for B recipients)
* Positive serology for human immunodeficiency virus (HIV)
* Clinical signs of hepatitis B virus (HBV) or hepatitis C virus (HCV) infections
* Clinical signs of cytomegalovirus (CMV) or Epstein-Barr virus (EBV) infections
* Positive test for severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) (according to local hospital routines)
* Active tuberculosis
* Severe other conditions requiring treatment and close monitoring, e.g. cardiac failure ≥grade 4 (New York Heart Association), unstable coronary disease or oxygen dependent chronic obstructive pulmonary disease (COPD)
* Any condition that in the view of the Investigator precludes transplantation
* History of a proven hypercoagulable condition
* Present or history of thrombotic thrombocytopenic purpura (TTP), or known familial history of TTP
* Intake of investigational drugs within 5 half-lives of the drug or 3 months, whichever is the longest
* Contemporaneous participation in a medical device study
* Known mental incapacity or language barriers precluding adequate understanding of the Informed Consent information and the trial activities
* Inability by the judgement of the investigator to participate in the trial for any other reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Mean estimated glomerular filtration rate (eGFR) at 12 months | 12 months after randomization
  eGFR is a measure of kidney function and will be compared between treatment arms.
  eGFR will be calculated based on p-creatinine according to the modification of diet in renal disease (MDRD) equation.
  eGFR for a kidney with normal function is 90 mL/min/1.73m2. Kidney disease is characterised by a decreased eGFR value. For randomized patients who do not undergo transplantation, lose their graft or die before 12 months, eGFR will be set to zero, consistent with kidney failure.

SECONDARY OUTCOMES:
Patient survival at 12 months | 12 months after randomization
  Patient survival will be summarized by end of trial and compared between treatment arms.

OTHER OUTCOMES:
Frequency of dialysis dependency at 12 months | 12 months after randomization
  Dialysis dependency is a measure of kidney function. A comparison between treatment arms will be done. Patients who are lost to follow up will be imputed as being dialysis-dependent.
Graft failure-free survival at 12 months | 12 months after randomization
  Graft failure-free survival is defined as the time from randomization to the first of either graft loss or death and will be compared between treatment arms.
Graft survival at 12 months | 12 months after randomization
  Graft survival will be compared between treatment arms in transplanted patients. Time to graft loss will be presented.
Frequency of wait-list categories at 12 months | 12 months after randomization
  Frequency of patients on different wait-list categories (i.e. on waitlist, temporarily delisted, delisted, dead) will be summarized by randomized treatment group
Frequency of delayed graft function | Within 7 days after transplantation
  Delayed graft function is defined as need for dialysis within 7 days of transplantation. Delayed graft function will be summarized by randomized treatment group
Antibody-mediated rejection (AMR) frequency | During 12 months after randomization
  Confirmed AMRs will be summarized by treatment. Presumed/suspected AMRs not confirmed with biopsies will be recorded as AE/SAE.
Cell-mediated rejection (CMR) frequency | During 12 months after randomization
  Confirmed CMRs will be summarized by treatment. Presumed/suspected CMRs not confirmed with biopsies will be recorded as AE/SAE.
Conversion of positive crossmatch test to negative | Within 4 hours after imlifidase treatment
  Imlifidase is highly efficacious in converting a positive crossmatch test to a negative. This outcome will be assessed for patients treated with imlifidase.
Donor specific antibody (DSA) levels for all antibodies with a mean fluorescence intensity (MFI) of ≥1000 | Prior first dose, 2, 4, 24, 48, 72 h and Days 5, 6, 8,15 and Months 1, 3, 6, 8, 10, and 12
  Analysis of DSAs will be done in serum from patients randomized to imlifidase using an IgG single antigen solid-phase immunoassay (SAB-HLA). Least square mean and standard error of DSA levels will be displayed over time.
Anti-drug antibodies (ADA) | Prior first dose, 48 hours, Days 8, 15, and Months 1, 2, 3, 6, 8, 10, and 12
  Immunogenicity towards imlifidase will be assessed by the measurement of ADA levels in patient serum using a customized ImmunoCAP analysis.
Imlifidase pharmacokinetics (AUC) | Within 24 hours prior to imlifidase treatment and up to Day 15
  AUC = Area under the imlifidase plasma concentration versus time curve
Imlifidase pharmacokinetics (Cmax) | Within 24 hours prior to imlifidase treatment and up to Day 15
  Cmax = Maximum observed plasma concentration of imlifidase following dosing
Imlifidase pharmacokinetics (tmax) | Within 24 hours prior to imlifidase treatment and up to Day 15
  tmax = Time point for maximum observed plasma concentration of imlifidase following dosing
Imlifidase pharmacokinetics (t1/2) | Within 24 hours prior to imlifidase treatment and up to Day 15
  t1/2 = Terminal half-life of imlifidase
Imlifidase pharmacokinetics (CL) | Within 24 hours prior to imlifidase treatment and up to Day 15
  CL = Clearance of imlifidase
Imlifidase pharmacokinetics (Vz) | Within 24 hours prior to imlifidase treatment and up to Day 15
  Vz = Apparent volume of distribution during terminal phase
Imlifidase pharmacodynamics | Within 24 hours prior to imlifidase treatment and up to Day 10
  Concentration of IgG in patient serum will be measured. Scoring of IgG fragments will be done.
Safety as measured by adverse events (AEs) | From signing informed consent to 12 months
  Safety is assessed as type, frequency and intensity of adverse events (AEs)/Serious adverse events (SAEs) including clinically relevant changes in clinical laboratory tests, vital signs and ECG)
Safety as measured by serious adverse events (SAEs) | From signing informed consent to 12 months
  Safety is assessed as type and frequency serious adverse events (SAEs)
Safety as measured by other adverse events (AEs) | From signing informed consent to 12 months
  Safety is assessed as type and frequency of other adverse events (AEs) - i.e. not including SAEs
Change in patient-reported life participation, as measured by PROMIS-SF-8a | At pre-screening and at 12 months after randomization
  The PROMIS Social Health domain "Ability to participate in social roles & activities PROMIS-SF-8" will be used as a measure of the patients' health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (25):
- United States (25):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Banner Health - University Medical Center - Phoenix, Phoenix, Arizona
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Keck Hospital of University of Southern California (USC), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sutter Health - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco (UCSF) Medical Center, San Francisco, California
  - Georgetown Transplant Institute, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - New York University (NYU) Langone Transplant Institute, NYU Langone Health, New York, New York
  - Columbia University, New York, New York
  - New York-Presbyterian - Weill Cornell Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Penn Medicine, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Methodist Hospital Specialty and Transplant, San Antonio, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No